CLINICAL TRIAL: NCT03436758
Title: Validation of Addition of Uterine Fluid to Human Embryo Culture Medium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IVI Murcia (Other)
Collaborators: Universidad de Murcia (Other)
Responsible Party: Sponsor
Other Study IDs: 1607-MUR-055-JL
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Infertility
Keywords: uterine fluids; Biobank; culture medium
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — uterine fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infertility or infertility affects about 15% of couples of reproductive age. It is estimated that 80 million people around the world suffer from this problem. Assisted reproduction techniques (ART) use culture media (during in vitro fertilization or early embryo development) with protein sources that are very different from natural sources. This media could produce an added stress to the gametes and embryos that could cause epigenetic alterations and health effects during adult life.

Our working hypothesis is based on studies in animal models (pig and cow), in which it was observed that the culture media with reproductive fluids used as additives instead of conventional sources of proteins (such as serum albumin) , produce embryos with an epigenetic profile closer to that of embryos generated in the maternal oviduct. Moreover, with these fluids, blastocysts obtained have a greater number of cells and hatchability than those produced with serum albumin alone.

Therefore, the University of Murcia, with an extensive experience in this area, and the IVI Murcia (Valencian Infertility Institute) research team have come together to launch this research project in order to determine the advantages of the use of human reproductive fluids as additives in embryonic culture media. To do this, 2 specific objectives are proposed,:

1. Creation of the first collection of human uterine fluid samples for Assisted Reproduction use.
2. To evaluate the use of uterine fluid as a media supplement in the culture media for assisted reproduction techniques, by evaluating embryo quality cultured with autologous fluid from voluntary patients (autologous culture)

This achievement would allow us the development of protocols in the nearest ART physiological conditions which represent not only a technical challenge but a biomedical responsibility that must be addressed to prevent future diseases of the offspring.

DETAILED DESCRIPTION:
1. Creation of the first collection of human uterine fluid samples for Assisted Reproduction use. Female reproductive system will be collected at the Virgen de la Arrixaca University Clinical Hospital from surgical pieces of patients undergoing surgical procedures. IVI Murcia Clinics uterine fluids from oocyte donors will be collected. These fluids will be store in the Arrixaca Hospital Biobank for future researches.
2. Validation of the addition of uterine fluid to human embryonic culture media:

Couples undergoing assited Reproduction Treatment in IVI Murcia will be asked for their inclusion in this study. Uterine fluid will be take 48 hours after peak of LH (luteinizing hormone), in natural cycle. Oocytes from these patients, will be divided into two groups: Half of the zygotes of each patient, control group, will be grown in the conditions usually used in the clinic, and the other half, experimental group, will add 1-5% of uterine fluid from the patient (v / v)

On day 3 and on day 5 of culture the quality of the embryos in both groups will be assessed according to the usual criteria of the clinic and the best quality and highest probability of implantation will be transferred, following the usual clinical practice. The samples of uterine fluid, after the initial processing in the IVI-Murcia clinic will be transferred to the Department of Physiology of the University of Murcia where they will be fractionated to perform a quality control according to the following specifications:

Uterine fluid pH 7.0-7.6 Osmolarity (mOsm / kg) 260-320 Endotoxin (EU / mL) <0.15 Sterility No growth

Only samples that meet these criteria will continue to be part of the study

ELIGIBILITY:
Inclusion Criteria:

* Couples in icsi treatment

Woman:

BMI between 17 and 30.Under controlled ovarian stimulation and at least 8 metaphase II oocytes collected

Man:

Sperm concentration higher than 5 million sperm / ml

Exclusion Criteria:

* Woman:

Diagnosis of endometriosis Uterine pathology that compromises embryonic development Patients undergoing treatment for repeat abortion or implantation failures Abnormal karyotype Patients included in the Pre-Implantation Genetic Diagnosis (DPI) program

Male:

Men whit abnormal karyotype, High values of DNA fragmentation Abnormal FISH (Fluorescence in situ Hybridization) Sperm from epididymal aspirate or testicular biopsy

Ages: 18 Years to 39 Years | Sex: All
Age Groups: Adult
Study Population: infertility couples
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
embryo quality | embryo quality will be analyze on day 3 and 5 after fertilization
  Number of embryo with A or B quality according to ASEBIR (Spanish association for the study of the biology of reproduction) criteria

SECONDARY OUTCOMES:
Pregnancy rate | between 14-16 days after fertilization
  serum levels of chorionic gonadotropin Beta (Beta-hCG)
ongoing pregnancy | 16-18 week after fertilization
  ultrasonography
implantation rate | 24 days after fertilization
  number of embryos implanted/number of embryos transferred x100
pregnancy loss rate | 10 days after B-hCG evaluation at end of pregnancy
  number of miscarriages/ number of ongoing pregnancy x100

CONTACTS AND LOCATIONS:
Overall Officials: Jose Landeras, MD, Principal Investigator — IVI-RMA
Locations (1):
- IVI Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coy P, Jimenez-Movilla M, Garcia-Vazquez FA, Mondejar I, Grullon L, Romar R. Oocytes use the plasminogen-plasmin system to remove supernumerary spermatozoa. Hum Reprod. 2012 Jul;27(7):1985-93. doi: 10.1093/humrep/des146. Epub 2012 May 3. PMID 22556378
- [Result] Aviles M, Gutierrez-Adan A, Coy P. Oviductal secretions: will they be key factors for the future ARTs? Mol Hum Reprod. 2010 Dec;16(12):896-906. doi: 10.1093/molehr/gaq056. Epub 2010 Jun 28. PMID 20584881
- [Result] Belva F, Bonduelle M, Roelants M, Michielsen D, Van Steirteghem A, Verheyen G, Tournaye H. Semen quality of young adult ICSI offspring: the first results. Hum Reprod. 2016 Dec;31(12):2811-2820. doi: 10.1093/humrep/dew245. Epub 2016 Oct 5. PMID 27707840
- [Result] Chiu PC, Chung MK, Koistinen R, Koistinen H, Seppala M, Ho PC, Ng EH, Lee KF, Yeung WS. Cumulus oophorus-associated glycodelin-C displaces sperm-bound glycodelin-A and -F and stimulates spermatozoa-zona pellucida binding. J Biol Chem. 2007 Feb 23;282(8):5378-88. doi: 10.1074/jbc.M607482200. Epub 2006 Dec 27. PMID 17192260
- [Result] Coy P, Canovas S, Mondejar I, Saavedra MD, Romar R, Grullon L, Matas C, Aviles M. Oviduct-specific glycoprotein and heparin modulate sperm-zona pellucida interaction during fertilization and contribute to the control of polyspermy. Proc Natl Acad Sci U S A. 2008 Oct 14;105(41):15809-14. doi: 10.1073/pnas.0804422105. Epub 2008 Oct 6. PMID 18838686
- [Result] Coy P, Grullon L, Canovas S, Romar R, Matas C, Aviles M. Hardening of the zona pellucida of unfertilized eggs can reduce polyspermic fertilization in the pig and cow. Reproduction. 2008 Jan;135(1):19-27. doi: 10.1530/REP-07-0280. PMID 18159080
- [Result] Gabler C, Chapman DA, Killian GJ. Expression and presence of osteopontin and integrins in the bovine oviduct during the oestrous cycle. Reproduction. 2003 Dec;126(6):721-9. PMID 14748691